CLINICAL TRIAL: NCT06195761
Title: Radiographic Assessment of Computer Guided Modified Ridge Splitting Technique Versus Conventional Free Hand Technique in Management of Horizontal Deficiency in Posterior Mandible: a Randomized Control Clinical Trial
Brief Title: Computer Guided Modified Ridge Splitting Versus Free Hand Technique in Horizontal Deficiency in Posterior Mandible
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina ElHadidi Sobhi Ramzi Michael, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: computer guided modified ridge
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Horizontal Bone Augmentation; Horizontal Ridge Deficiency
Keywords: computer guided modified ridge splitting; computer guided modified cortical shell technique; guided modified ridge splitting in posterior mandible

STUDY DESIGN:
Intervention Model Description: treatment plan includes harvesting and fixing the bone graft in posterior mandibular area using a computer-modified surgical guide
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided modified ridge splitting technique (study group) (Experimental): The first treatment plan includes harvesting and fixing the bone graft in posterior mandibular area using a computer-modified surgical guide.
  Interventions: Procedure: computer guided modified ridge splitting technique in horizontal bone deficiency in posterior mandible
- conventional modified ridge splitting technique (control group) (Experimental): The second treatment plan includes manually harvesting and fixing the bone graft in posterior mandibular area without a surgical guide
  Interventions: Procedure: free hand modified ridge splitting technique in horizontal bone deficiency in posterior mandible

INTERVENTIONS:
Procedure: computer guided modified ridge splitting technique in horizontal bone deficiency in posterior mandible — treatment plan includes harvesting and fixing the bone graft in posterior mandibular area using a computer-modified surgical guide
  Other Names: computer guided modified cortical shell technique
  Arms: computer guided modified ridge splitting technique (study group)
Procedure: free hand modified ridge splitting technique in horizontal bone deficiency in posterior mandible — treatment plan includes manually harvesting and fixing the bone graft in posterior mandibular area without a surgical guide.
  Other Names: conventional modified cortical shell technique
  Arms: conventional modified ridge splitting technique (control group)

SUMMARY:
To assess the accuracy of the computer assessed guides in horizontal bone augmentation achieved at posterior mandible using guided modified ridge splitting technique versus free hand modified ridge splitting technique

DETAILED DESCRIPTION:
The first treatment plan includes harvesting and fixing the bone graft in posterior mandibular area using a computer-modified surgical guide.

The second treatment plan includes manually harvesting and fixing the bone graft in posterior mandibular area without a surgical guide.

ELIGIBILITY:
Inclusion Criteria:

* posterior mandible with horizontal deficient alveolar ridge that is from 2 to 4 mm measured from the crest of the alveolar ridge buccolingually
* Age range from 25-55 years. No sex predilection.
* Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* Patients of adequate alveolar bone width.
* Both genders males and females will be included
* Normal vertical dimension with normal inter-arch space. The minimum number of missing teeth in the posterior mandible alveolar ridge is two adjacent anterior teeth

Exclusion Criteria:

* Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.
* Previous grafting procedures in the edentulous area.
* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Immunosuppressed or immunocompromised
* Heavy smokers
* Patients undergo medication interfere with bone healing

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Computer Assessed Guide in the study group | immediately postoperative
  Accuracy of the Computer Assessed Guide in the study group In comparison with the control group between predicted and immediately postoperative horizontal bone width with Cone beam computed tomography in Millimeters measurement tool is CBCT scan superimposition in mm

SECONDARY OUTCOMES:
Alveolar ridge horizontal bone gain | 4 months
  measure the amount of horizontal bone width gaining by postoperative cone beam computed tomography in millimeters measurement tool is CBCT scan superimposition in mm

OTHER OUTCOMES:
soft tissue dehiscience | 2 months postoperatively
  measument tool is periodontal probe to measure the amount of dehscience of the soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mounir Shaker, BDS,MSc,PHD, Study Chair — Cairo University; Rofaida Atef Abaas, BDS,MSc,PHD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Manial, Egypt

REFERENCES:
- [Result] Al-Ani O, Nambiar P, Ha KO, Ngeow WC. Safe zone for bone harvesting from the interforaminal region of the mandible. Clin Oral Implants Res. 2013 Aug;24 Suppl A100:115-21. doi: 10.1111/j.1600-0501.2011.02393.x. Epub 2012 Jan 11. PMID 22233422
- [Result] Sanchez-Labrador L, Molinero-Mourelle P, Perez-Gonzalez F, Saez-Alcaide LM, Brinkmann JC, Martinez JL, Martinez-Gonzalez JM. Clinical performance of alveolar ridge augmentation with xenogeneic bone block grafts versus autogenous bone block grafts. A systematic review. J Stomatol Oral Maxillofac Surg. 2021 Jun;122(3):293-302. doi: 10.1016/j.jormas.2020.10.009. Epub 2020 Nov 5. PMID 33161168
- [Result] De Stavola L, Fincato A, Bressan E, Gobbato L. Results of Computer-Guided Bone Block Harvesting from the Mandible: A Case Series. Int J Periodontics Restorative Dent. 2017 Jan/Feb;37(1):e111-e119. doi: 10.11607/prd.2721. PMID 27977816
- [Result] Schwartz-Arad D, Levin L, Sigal L. Surgical success of intraoral autogenous block onlay bone grafting for alveolar ridge augmentation. Implant Dent. 2005 Jun;14(2):131-8. doi: 10.1097/01.id.0000165031.33190.0d. PMID 15968184
- [Result] Assaf A, Saad M, Daas M, Abdallah J, Abdallah R. Use of narrow-diameter implants in the posterior jaw: a systematic review. Implant Dent. 2015 Jun;24(3):294-306. doi: 10.1097/ID.0000000000000238. PMID 25851960